CLINICAL TRIAL: NCT02790047
Title: Effect of Home-base Exercise Program With a Conical Positive Expiratory Pressure Device on Physical Performance and Health Related Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Home-base Exercise With Conical-PEP Device on Physical Performance and Quality of Life in COPD
Acronym: HBEcPEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Chatchai Phimphasak, Principal Investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHD/0082/2556
Record Dates: First submitted 2016-02-02; First posted 2016-06-03 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Exercise Therapy; Positive Expiratory Pressure; Physical Fitness; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-base exercise (Active Comparator): Patients will receive intervention as following
  1. A home-base exercise program
  2. Health education
  3. Breathing strategies for self secretion clearance
  4. The medication following the COPD GOLD guidelines (2015)
  Interventions: Other: A home-base exercise program; Other: Health education; Other: ฺBreathing strategies for self secretion clearance; Drug: The medication following the COPD GOLD guidelines (2015)
- Home-base exercise with a PEP mask (Experimental): Patients will receive intervention as following
  1. A home-base exercise program with using a non-re-breathing face mask with conical-PEP device during an interval endurance spot marching exercise
  2. Health education
  3. Breathing strategies for self secretion clearance
  4. The medication following the COPD GOLD guidelines (2015)
  Interventions: Device: A non-re-breathing face mask with conical-PEP device; Other: A home-base exercise program; Other: Health education; Other: ฺBreathing strategies for self secretion clearance; Drug: The medication following the COPD GOLD guidelines (2015)

INTERVENTIONS:
Device: A non-re-breathing face mask with conical-PEP device — Participant will use a non-re-breathing face mask with conical-PEP device during an interval endurance spot marching exercise.
  Arms: Home-base exercise with a PEP mask
Other: A home-base exercise program — Duration of the program is 8 weeks A frequency of exercise session is 3 to 5 sessions per week A content of each exercise session includes
  1. Stretching exercise (shoulder, trunk and leg muscles) to warm up for 5 to 10 minutes
  2. Interval endurance exercise using a spot marching movement for 30 to 40 minutes. In each phase of spot marching exercise, patients will perform the exercise from 0 to 3 or 4 score of 10 score of a modified dyspnea Borg scale, they will record exercise the exercise duration time. Then, they will be required to rest until a modified dyspnea Borg scale < 1 score. Next, they will perform the next interval of spot marching exercise with the same protocol.
  3. Stretching exercise (shoulder, trunk and leg muscles) to cool down for 5 to 10 minutes
Other: Health education — Health education include
  1. Knowledge of COPD disease
  2. Smoking status and smoking cessation
  3. Medication correctly
  4. Self dyspnea management
  5. Basic nutrition for COPD
Other: ฺBreathing strategies for self secretion clearance — Using a modified active cycle breathing technique (mACBT) include
  1. Control breathing
  2. Pursed lip breathing (PLB)
  3. Slow inhale with sustain thoracic expansion for 3 sec and exhale with PLB technique
  4. Force expiratory technique (FET) with low to medium lung volume
  5. Huffing or coughing
Drug: The medication following the COPD GOLD guidelines (2015) — Patients will receive medications following the COPD GOLD guidelines (2015). The medication names were listed below
  1. Bata 2 agonist (short acting); Salbutamol (oral or inhaler), Terbutaline (oral)
  2. Bata 2 agonist (long acting); Bambuterol (oral), Procaterol (oral), Salmeterol (inhaler), Formoterol (inhaler)
  3. Xanthine derivative (sustained release theophylline)
  4. Anticholinergic; Tiotropium(inhaler), Ipratropium bromide (inhaler)
  5. Corticosteroids; Beclomethasone (inhaler), Budesonide(inhaler), Fluticasone(inhaler)
  6. Combined anticholinergic+ Beta 2-agonist; Ipratropium+fenoterol (inhaler), Ipratropium+salbutamol (inhaler)
  7. Combined Beta 2-agonist+ corticosteroids; Formoterol+ Budesonide(inhaler), Salmeterol+ Fluticasone(inhaler)

SUMMARY:
The aim of this study to investigate the efficacy of a home-base exercise program with a new conical PEP device on physical performance and health related quality of life in COPD patients.

DETAILED DESCRIPTION:
The key pathophysiology of COPD is expiratory flow limit and hyperinflation that is a major factor related exertional dyspnea and exercise limitation. When expiratory minute volume( V ̇E) raise up while exercise, respiratory response by increase respiratory rate (RR) and tidal volume (VT), force exhalation occur lead to develop premature airway closer. These generate dynamic air tapping breath by breath and result in dynamic hyperinflation (DH). The DH limits VT expansion, increase respiratory muscle load, and it is a major cause related dyspnea and exercise termination. Furthermore, Pre-inflammatory products from the COPD lung contribute to another system, and provoke systemic inflammation lead to nutritional abnormalities, weight loss, skeletal muscle dysfunction, osteo-skeletal effect, cardiovascular effect and psychological effect. All of these affect the exercise tolerance and gradually affect physical activity and health-related quality of life (HRQL) as well.

COPD GOLD guideline states that goal for treatments of stable COPD comprise of relive symptoms, improve exercise tolerance, improve health status, prevent disease progression and reduce mortality. Several evidences have suggested an effect of pulmonary rehabilitation (PR) in patient with stable COPD and following acute exacerbation. Strong evidences reported that the PR program could improve exercise tolerance, reduce dyspnea, decrease fatigue and improve health-related quality of life.

The core stone of PR is an exercise program. Several types of exercise were published such as endurance exercise, interval exercise, strengthening exercise, respiratory muscle strengthening and breathing exercise. Most COPD patient stop exercise causes from dyspnea that related DH development during exercise. Previous studies reported various strategies to reduce DH development during exercise for extending exercise time or increase exercise capacity in immediate effect such as bronchodilators , hyperoxic breathing, heliox breathing, positive pressure therapy by non-invasive positive pressure ventilation (NIPPV), by pursed lip breathing (PLB) and by positive expiratory pressure (PEP) device.

The PEP therapy have been conventionally using for reduce premature airway closer by moving equal pressure point from distal to proximal, improve gas exchange and improve secretion clearance. In the past decade, the knowledge of dynamic hyperinflation in COPD patient has rapidly glowed up. The PEP device and PLB have used to reduce DH development during exercise that reported in only 5 studies. They expected that delay DH development, it may delay exertional dyspnea, and may result in improve exercise capacity.

Three studies reported DH parameter at pre and post exercise. Results indicated that using the PEP device can reduce DH when measuring immediate post exercise. However, effects of positive pressure therapy (PEP device and PLB) on exercise capacity were also inconclusive. But three studies showed positive effect of PEP therapy on exercise capacity.

Training effect of PEP therapy on physical performance and quality of life was present in two studies. The first study showed the benefit of breathing retraining (including PLB, and other breathing techniques) that were integrated to all daily activities and exercise program, superior than control group in peak oxygen consumption after 7th week of exercise program. The second study applied PLB to reduce DH during exercise program. They found that after ten sessions (within 3 to 4 weeks) of program, both PLB and control groups significantly improve 6 minute walk distance and quality of life, but non-significant effect between groups. To date there was only two studies of PEP therapy applying to exercise program, and results were not conclusive.

In spite of the PLB was wildly used, but positive pressure from this technique was reported about 5 cm H2O, it is lower boundary of therapeutic pressure range (5 to 20 cm H2O), this may result in a non-success of DH reduction. Consequently, The PEP device may be a convenient alternative way to generate positive pressure within therapeutic range for reduces DH during exercise or daily activities living. This may increase patient's physical performance and quality of life greater that exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (with FEV1 ≤70% predicted)

Exclusion Criteria:

* Exacerbate within a month prior, which was a cause of admission to the hospital emergency room or been admitted to hospital.
* Are changed medicines within a month ago.
* Have been used home oxygen therapy.
* Have musculoskeletal or neuromuscular problem affecting balance and walking. and spot marching exercise.
* Using walking aid device.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change of 6 minute walk distance (6MWD) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The 6MWD represents physical performance of COPD pateints.

SECONDARY OUTCOMES:
Change of St George's Respiratory Questionnaire (SGRQ) score | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The SGRQ represents health related quality of life of COPD patients.
Incremental sport marching exercise test (ISMT) | baseline
  The ISMT is combination movement of high arm and leg raising on the spot . Patient will start ISMT with 60 or 70 steps/minute and increase 10 to 20 steps/minute every 2 minutes until symptom limited. Aim of this test is to fine maximum step rate and step rate which patient perceive at least moderate dyspnea or breathlessness. The proper step rate will use in endurance spot marching exercise test (ESMT).
Change of endurance exercise time of endurance sport marching exercise test (ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The ESMT is a physical performance parameter. The exercise capacity of this test is endurance exercise time. Patents will perform ESMT with constant step rate until symptom limit or exercise time up to 25 minute.
Change of resting inspiratory capacity (IC) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The resting IC reflects static hyperinflation.
Change of end exercise inspiratory capacity in ESMT (IC-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The end exercise IC reflects dynamic hyperinflation. patient will be measured the end exercise IC at immediate post ESMT.
Change of resting slow vital capacity (SVC) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The resting SVC reflect static hyperinflation
Change of end exercise slow vital capacity in ESMT (SVC-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The resting SVC reflect dynamic hyperinflation.patient will be measured the end exercise IC at immediate post ESMT.
Change of resting heart rate (HR) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting EKG for 20 minutes. the EKG will be analysis to resting HR
Change of resting respiratory rate (RR) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting RR for 20 minutes. The RR will be recorded every minute.
Change of resting pulse oxygen saturation (SpO2) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting SpO2 for 20 minutes. The SpO2 will be recorded every minute.
Change of resting end tidal carbon dioxide (PetCO2) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting PetCO2 for 20 minutes. The PetCO2 will be recorded every minute.
Change of resting systolic blood pressure (SBP) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting SBP every 2 minutes for 20 minutes.
Change of resting diastolic blood pressure (DBP) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting DBP every 2 minutes for 20 minutes.
Change of resting mean arterial pressure (MAP) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting MAP every 2 minutes for 20 minutes.
Change of resting pusle wave velocity (PWV) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be continuously measured resting EKG and photoplethysmography (PPG) for 20 minutes. The pulse transit time will be collected from EKG and PPG, then the pulse transit time in each patient will divide by a length of their arm (from jugular notch to tip of index finger )
Change of end exercise heart rate in ESMT (HR-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be continuously measured EKG during ESMT. The investigators will collect end exercise HR at immediate post ESMT and every minute in recovery period for 10 minutes.
Change of end exercise rating perceive of breathlessness in ESMT (RPB-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will rate their breathlessness using 10 scale of modified Borg dyspnea scale at pre-ESMT, during ESMT every minute, end ESMT and every minute in recovery period for 10 minute.
Change of end exercise respiratory rate in ESMT (RR-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded RR at pre-ESMT, during ESMT every minute, end ESMT and every minute in recovery period for 10 minutes.
Change of end exercise tidal volume in ESMT (RR-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded tidal volume at pre-ESMT, end ESMT and end recovery period for 10 minutes.
Change of end exercise minute ventilation in ESMT (RR-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded minute ventilation at pre-ESMT, end ESMT and end recovery period for 10 minutes.
Change of end exercise pulse oxygen saturation in ESMT (SpO2-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded SpO2 at pre-ESMT, during ESMT every minute, end ESMT and every minute in recovery period for 10 minutes.
Change of end exercise end tidal carbon dioxide in ESMT (PetCO2-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded PetCO2 at pre-ESMT, during ESMT every minute, end ESMT and every minute in recovery period for 10 minutes.
Change of end exercise systolic blood pressure in ESMT (SBP-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded SBP at pre-ESMT, immediate end ESMT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise diastolic blood pressure in ESMT (DBP-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded DBP at pre-ESMT, immediate end ESMT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise mean arterial pressure in ESMT (MAP-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded MAP at pre-ESMT, immediate end ESMT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise pulse wave velocity in ESMT (PWV-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be continuously measured EKG and photoplethysmography (PPG) at pre ESMT during ESMT and recovery period for 10 minutes. The pulse transit time will be collected from EKG and PPG at end of ESMT, then the pulse transit time in each patient will divide by a length of their arm (from jugular notch to tip of index finger )
Change of end exercise leg fatigue score in ESMT (LEG-ESMT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will rate their leg fatigue using 10 scale of modified Borg leg fatigue scale at pre-ESMT, during ESMT every minute, end ESMT and every minute in recovery period for 10 minute.
Change of end exercise heart rate in 6MWT (HR-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be continuously measured HR during 6MWT. The investigators will collect end exercise HR at immediate post 6MWT and every minute in recovery period for 10 minutes.
Change of end exercise rating perceive of breathlessness in 6MWT (RPB-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will rate their breathlessness using 10 scale of modified Borg dyspnea scale at pre-6MWT, during 6MWT every minute, end 6MWT and every minute in recovery period for 10 minute.
Change of end exercise respiratory rate in 6MWT (RR-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded RR at pre-6MWT, during 6MWT every minute, end 6MWT and every minute in recovery period for 10 minutes.
Change of end exercise pulse oxygen saturation in 6MWT (SpO2-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded SpO2 at pre-6MWT, during 6MWT every minute, end 6MWT and every minute in recovery period for 10 minutes.
Change of end exercise end tidal carbon dioxide in 6MWT (PetCO2-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded PetCO2 at pre-6MWT, during 6MWT every minute, end 6MWT and every minute in recovery period for 10 minutes.
Change of end exercise systolic blood pressure in 6MWT (SBP-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded SBP at pre-6MWT, immediate end 6MWT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise diastolic blood pressure in 6MWT (DBP-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded DBP at pre-6MWT, immediate end 6MWT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise mean arterial pressure in 6MWT (MAP-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be recorded MAP at pre-6MWT, immediate end 6MWT and every 2 minutes in recovery period for 10 minutes.
Change of end exercise leg fatigue score in 6MWT (LEG-6MWT) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will rate their leg fatigue using 10 scale of modified Borg leg fatigue scale at pre-6MWT, during 6MWT every minute, end 6MWT and every minute in recovery period for 10 minute.
Change of resting heart rate variability (HRV) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will be measured resting EKG for 20 minutes. The EKG will be analysis to HRV
Change of Chronic Obstructive Pulmonary Disease Assessment Test (CAT) score | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The CAT is health related quality of life questionnaire.
Change of Modified Medical Research Council Questionnaire (mMRC) score | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The mMRC is one of dyspnea parameters. It is ordinal data.
Change of hand grip force | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The hand grip force represents general health status of patients. patient will be assessed both dominated and non-dominated hands.
Change of force vital capacity (FVC) and force vital capacity %predicted | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  patient will perform spirometry in FVC maneuver to record post bronco-dilator force vital capacity following American Thoracic Society (ATS) /European Respiratory Society (ERS) statement for spirometry (2005).
Change of force expiratory volume in one second (FEV1) and FEV1%predicted | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  patient will perform spirometry in FVC maneuver to record post bronco-dilator FEV1 following ATS/ERS statement for spirometry (2005).
Change of FEV1/FVC ratio | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  patient will perform spirometry in FVC maneuver to record post bronco-dilator FEV1/FVC ratio following ATS/ERS statement for spirometry (2005).
Change of peak expiratory flow rate (PEF) and PEF%predicted | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  patient will perform spirometry in FVC maneuver to record post bronco-dilator PEF following ATS/ERS statement for spirometry (2005).
Change of Maximum inspiratory pressure (MIP) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will maximum inhale as fast as possible from functional residual capacity (FRC) to total lung capacity (TLC).
Change of Maximum expiratory pressure (MEP) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patients will maximum exhale as fast as possible from TLC to residual volume (RV).
Change of Baseline Dyspnea Index (BDI) | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The BDI is one of dyspnea parameters (questionnaire). Three dimension questions include; 1.effect of daily function on dyspnea, 2. effect of magnitude of task on dyspnea and 3. effect of magnitude off effort on dyspnea.
Change of Transition Dyspnea Index (TDI) | post home-base exercise program at 8th weeks and follow up at 5th months
  The TDI assesses change of dyspnea perception from the BDI in each dimensions. Patient will rate score from -6 to +6 (positive score reflect improve of dyspnea and negative score reflect worse dyspnea).
Change of number of step per day | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  The number of step per day represents physical activity using a pedometer. Patient will contact the pedometer from early wake up to go to bed with 10 day hours for 14 day before starting the home-base exercise program, post the home-base exercise program and 5th months . The researcher will record the regular step per day for 7 days to analysis.
Change of rate of using short acting bronco-dilator per week | baseline, post home-base exercise program at 8th weeks and follow up at 5th months
  Patient will be collected the rate of using short acting bronco-dilator per week as 2 months ago of the time frame.
Number of exacerbation event | Collecting from starting the homes-base exercise program to 5th months follow up.
  Definition of exacerbation is a cause of admission to the hospital emergency room or admitting to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Chulee U Jones, Ph.D., PT, Study Director — Khon Kaen University; Chatchai Phimphasak, M.Sc, PT, Principal Investigator — Khon Kaen University
Locations (2):
- Thailand (2):
  - School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen, Changwat Khon Kaen
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen

IPD SHARING:
Plan to Share IPD: Undecided